CLINICAL TRIAL: NCT03238742
Title: The Efficacy of Xuebijing Injection in Adult Patients With Sepsis
Brief Title: The Efficacy of Xuebijing Injection on Sepsis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southeast University, China (Other)
Collaborators: National Health and Family Planning Commission, P.R.China (Other Government)
Responsible Party: Principal Investigator, Songqiao Liu, Principle investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017ZDSYLL025-P01
Record Dates: First submitted 2017-07-29; First posted 2017-08-03 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Sepsis
Keywords: Xuebijing Injection, morality, sepsis
MeSH Terms: conditions — Sepsis | interventions — Xuebijing; Saline Solution

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blind (Participant, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): 100ml Xuebijing Injection will be dissolved in 100 mL of normal saline every 12 hours for 5 days in blind fashion.
  Interventions: Drug: Xuebijing Injection
- Placebo group (Placebo Comparator): normal saline 200 mL every 12 hours for 5 days
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Xuebijing Injection — 100ml Xuebijing Injection every 12 hours for 5 days
  Arms: Intervention Group
Drug: normal saline — 200ml normal saline every 12 hours for 5 days
  Other Names: NS
  Arms: Placebo group

SUMMARY:
The Efficacy of Xuebijing Injection in Adult Patients with Sepsis

DETAILED DESCRIPTION:
The purpose of this placebo-controlled study is to determine if Xuebijing Injection treatment provides significant mortality reduction improvement in patients with sepsis compared with placebo treatment in patients receiving the current standard of care for sepsis. This study will also assess the effectiveness of Xuebijing Injection in reducing 28-day mortality in patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for inclusion if all of the inclusion criteria are met

1. Sepsis-3 criteria from Society of Critical Care Medicine (SCCM) /European Society of Intensive Care Medicine (ESICM)
2. 18≤ age ≤75years
3. 2 ≤SOFA ≤13
4. obtain informed consent

Exclusion Criteria:

1. Diagnosis of sepsis for more than 48 h;
2. Pregnant and lactating women;
3. Severe primary disease including unrespectable tumours, blood diseases and Human Immunodeficiency Virus (HIV);
4. Severe liver and kidney dysfunction (single liver or kidney SOFA score ≥ 3 points);
5. Use of an immunosuppressant or having an organ transplant within the previous 6 months;
6. Participating in other clinical trials in the previous 30 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1817 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2019-07-28 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 28 Days after randomization
  Death from all causes at 28-days

SECONDARY OUTCOMES:
Death in ICU | 28 Days after randomization
  Death from all causes at ICU discharge
SOFA score | Day 0,3,6 after randomization
  Total Sequential Organ Failure Assessment (SOFA) score(0-24) ，higher values represent a worse outcome
APACHEⅡ | Day 0,3,6 after randomization
  Acute Physiology and Chronic Health Evaluation (include Acute physiology score, APS and age and Chronic physiology score, totally 0-71 Points)
Duration of mechanical ventilation | 28 days after randomization
  Duration of mechanical ventilation in ICU
ICU stay | 28 days after randomization
  Duration of stay in ICU
Concentration of C-reactive protein | 0,3,6days after randomization
  C-reactive protein at 0, 3,6 days after randomization
Concentration of Procalcitonin | 0,3,6 days after randomization
  Procalcitonin at 0,3,6days after randomization
Percentage of Human Leukocyte Antigen-DR | 0，6 days after randomization
  Human Leukocyte Antigen-DR at 0, 6 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Qiu Haibo, Dr., Principal Investigator — Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Mortality
Supporting Information: Study Protocol
Time Frame: Study published
Access Criteria: Supplyment

REFERENCES:
- [Derived] Lou X, Chen H, Shi N, Yu R, Li S, Yang Y, Liu S, Xie J, Qiu H. Treatment effects of Xuebijing injection in patients with sepsis by clinical phenotype: a post hoc analysis of the EXIT-SEP trial. EClinicalMedicine. 2025 Jul 9;86:103341. doi: 10.1016/j.eclinm.2025.103341. eCollection 2025 Aug. PMID 40666169
- [Derived] Liu S, Yao C, Xie J, Liu H, Wang H, Lin Z, Qin B, Wang D, Lu W, Ma X, Liu Y, Liu L, Zhang C, Xu L, Zheng R, Zhou F, Liu Z, Zhang G, Zhou L, Liu J, Fei A, Zhang G, Zhu Y, Qian K, Wang R, Liang Y, Duan M, Wu D, Sun R, Wang Y, Zhang X, Cao Q, Yang M, Jin M, Song Y, Huang L, Zhou F, Chen D, Liang Q, Qian C, Tang Z, Zhang Z, Feng Q, Peng Z, Sun R, Song Z, Sun Y, Chai Y, Zhou L, Cheng C, Li L, Yan X, Zhang J, Huang Y, Guo F, Li C, Yang Y, Shang H, Qiu H; EXIT-SEP Investigators. Effect of an Herbal-Based Injection on 28-Day Mortality in Patients With Sepsis: The EXIT-SEP Randomized Clinical Trial. JAMA Intern Med. 2023 Jul 1;183(7):647-655. doi: 10.1001/jamainternmed.2023.0780. PMID 37126332
- [Derived] Liu S, Yao C, Zhang J, Yang Y, Qiu H; EXIT-SEP Investigators. Efficacy of Xuebijing Injection for Sepsis (EXIT-SEP): protocol for a randomised controlled trial. BMJ Open. 2019 Aug 28;9(8):e028664. doi: 10.1136/bmjopen-2018-028664. PMID 31467049
- Available data/document: Clinical Review& Education: 2 — http://www.ncbi.nlm.nih.gov/pubmed/26903338 — Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC.The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016;315(8):801-10.